CLINICAL TRIAL: NCT01076348
Title: Medtronic Model 4965 Capsure Epi® Steroid-eluting Unipolar Epicardial Pacing Lead Post Approval Study
Brief Title: Model 4965 Post-Approval Study
Status: Completed | Type: Observational
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: 4965
Record Dates: First submitted 2010-02-24; First posted 2010-02-26 (Estimated); Results first posted 2012-08-23 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure; Pacing; Bradycardia; Arrhythmia
Keywords: Epicardial; Pacing Lead
MeSH Terms: conditions — Heart Failure; Bradycardia; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Safety and effectiveness will be summarized for the model 4965 lead. This study was conducted within Medtronic's System Longevity Study (SLS).

DETAILED DESCRIPTION:
As part of the requirement to satisfy the PMA Conditions of Approval for the Medtronic Model 4965 CapSure Epi® Steroid-Eluting Unipolar Epicardial Pacing Lead, 50 adult subjects who were ≥19 years old at time of implant were followed for one-year post-implant.

ELIGIBILITY:
Inclusion Criteria:

* Subjects or appropriate legal guardians provide written informed consent and/or authorization for access to and use of health information, as required by an institution's IRB/MEC/REB

AND one of the following (A, B, or C) must also apply:

A. Subjects indicated for implant or within six months post-implant of a Medtronic market-released lead connected to a market-released IPG, ICD, or CRT Device. The Medtronic lead must be used for a pacing, sensing, or defibrillation application.

B. Subjects who participated in a qualifying study of a Medtronic cardiac therapy product and for whom:

* product is market-released
* complete implant and follow-up data, including product-related adverse events, are available
* subject or appropriate legal guardian authorizes release of subject study data to SLS C. Subjects implanted with Medtronic CapSure Epi Leads (model 4965 and 4968) at a minimum of three pre-selected sites to retrospectively collect data for post approval requirements. Post approval requirements indicate 50 adult subjects implanted with a model 4965 and 100 subjects (pediatric and adult) implanted with a model 4968. The study plans to enroll approximately 100 subjects with a model 4965 lead and approximately 200 subjects with a model 4968 lead.

Note: Subjects currently active in the Chronic Lead Study or Tachyarrhythmia Chronic Systems Study will continue in the follow-up phase of the SLS.

Exclusion Criteria:

* Subjects receiving an implant of a Medtronic lead at a non-participating center and the implant data and current status cannot be confirmed within 30 days after implant
* Subjects who are, or will be inaccessible for follow-up at a SLS center
* Subjects implanted with a Medtronic cardiac therapy device whose predetermined enrollment limit for that specific product has been exceeded
* Subjects with exclusion criteria required by local law (EMEA only)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects 19 years or older implanted with Model 4965 Capsure Epi Lead.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 1996-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: 4965 Post-Approval Study Clinical Trial Leader, Study Chair — Medtronic
Locations (107):
- United States (84):
  - Birmingham, Alabama
  - Anchorage, Alaska
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Little Rock, Arkansas
  - Bakersfield, California
  - Chula Vista, California
  - Downey, California
  - East Palo Alto, California
  - Los Angeles, California
  - Salinas, California
  - Torrance, California
  - Van Nuys, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Clearwater, Florida
  - Jacksonville, Florida
  - Melbourne, Florida
  - Ocala, Florida
  - Wellington, Florida
  - Atlanta, Georgia
  - Columbus, Georgia
  - Marietta, Georgia
  - Oak Lawn, Illinois
  - Indianapolis, Indiana
  - Newburgh, Indiana
  - Des Moines, Iowa
  - Kansas City, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Alexandria, Louisiana
  - Baton Rouge, Louisiana
  - Salisbury, Maryland
  - Silver Spring, Maryland
  - Towson, Maryland
  - Grand Blanc, Michigan
  - Marquette, Michigan
  - Saginaw, Michigan
  - Southfield, Michigan
  - Robbinsdale, Minnesota
  - Rochester, Minnesota
  - Saint Paul, Minnesota
  - Kansas City, Missouri
  - Lebanon, New Hampshire
  - Browns Mills, New Jersey
  - Newark, New Jersey
  - Ocean City, New Jersey
  - Parlin, New Jersey
  - West Orange, New Jersey
  - Albuquerque, New Mexico
  - Mineola, New York
  - Rochester, New York
  - Greensboro, North Carolina
  - Hickory, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Toledo, Ohio
  - Portland, Oregon
  - Doylestown, Pennsylvania
  - Lancaster, Pennsylvania
  - Sayre, Pennsylvania
  - Columbia, South Carolina
  - Florence, South Carolina
  - Sioux Falls, South Dakota
  - Chattanooga, Tennessee
  - Germantown, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Amarillo, Texas
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - San Antonio, Texas
  - The Woodlands, Texas
  - Burlington, Vermont
  - Chesapeake, Virginia
  - Fairfax, Virginia
  - Olympia, Washington
  - Spokane, Washington
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Bedford Park, South Australia, Australia
- Austria (2):
  - Linz
  - Vienna
- Hasselt, Belgium
- Canada (7):
  - Calgary, Alberta
  - Hamilton, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Ste-Foy, Quebec
  - Regina, Saskatchewan
- Copenhagen, Denmark
- Marseille, France
- Homburg/Saar, Germany
- Italy (3):
  - Catanzaro
  - Reggio Emilia
  - Udine
- Netherlands (2):
  - Eindhoven
  - Rotterdam
- Belgrade, Serbia
- Valencia, Spain
- Skövde, Sweden
- Zurich, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study utilized centers that had implanted model 4965 leads in adult subjects to obtain information regarding safety, lead events, and lead survival.
Groups:
- Medtronic 4965 Subjects: Single arm registry of Model 4965 implanted patients
Period: Overall Study
Arm/Group | Medtronic 4965 Subjects
Started | 73
Completed | 51
Not Completed | 22

BASELINE CHARACTERISTICS:
Arm/Group | Medtronic 4965 Subjects
Number analyzed (Participants) | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 44
Region of Enrollment [Number; unit: participants]
  United States | 72
  Germany | 1

OUTCOME MEASURES:

1. Primary Outcome: Model 4965 Complication Free Rate
Description: A 4965 lead-related complication is an adverse event requiring invasive intervention to resolve. The complication-free rate is based on the number of leads analyzed.
Time Frame: 1 year
Population: Patients ≥ 19 yrs at implant of MDT 4965 Epicardial Lead.
Measure: Number (95% Confidence Interval); unit: Model 4965 complication free rate
Units Other Than Participants: 4965 leads
Groups:
- Medtronic 4965 Epicardial Lead: Subjects who were implanted with at least 1 model 4965 lead.
Arm/Group | Medtronic 4965 Epicardial Lead
Number analyzed (Participants) | 73
Number analyzed (4965 leads) | 98
Model 4965 complication free rate | 98.8 [91.8 to 99.8]

ADVERSE EVENTS:
Description: For this study, "serious" is defined as requiring an invasive intervention to resolve.
Arm/Group | Medtronic 4965 Subjects
Serious Adverse Events (participants affected / at risk) | 2/73
Other Adverse Events (participants affected / at risk) | 0/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medtronic 4965 Subjects (N=73)
Failure to capture (Vascular disorders) | 1 (1) — Intermittent
Lead conductor fracture (Vascular disorders) | 1 (1) — Lead electrically abandoned

LIMITATIONS AND CAVEATS:
The study cohort was limited to subjects >19 years of age at the time of implant, limiting the survival analysis of the Model 4965 lead in a pediatric population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No